CLINICAL TRIAL: NCT02954757
Title: Therapeutic Efficacy of High-intensity Focused Ultrasound in the Treatment of Uterine Adenomyosis
Brief Title: High-intensity Focused Ultrasound in Treatment of Uterine Adenomyosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Vincent YT Cheung, Dr., Queen Mary Hospital, Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW16-283
Record Dates: First submitted 2016-10-20; First posted 2016-11-03 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Adenomyosis
Keywords: uterine adenomyosis
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment arm (Experimental): HIFU treatment
  Interventions: Procedure: HIFU treatment

INTERVENTIONS:
Procedure: HIFU treatment — High intensity focused ultrasound

SUMMARY:
Uterine adenomyosis is a common uterine benign condition. They can cause abnormal menstrual bleeding, and menstrual pain. Although surgical intervention is the definitive treatment, some women prefer to have their uterus preserved. High-intensity focused ultrasound (HIFU) therapy is receiving increasing interest in the management of uterine adenomyosis by inducing focal thermocoagulation of the fibroids. Results obtained by various research groups have shown that HIFU treatment is safe, effective and is highly acceptable to patients. The main objective of this study is to evaluate the therapeutic efficacy of HIFU in the treatment of uterine adenomyosis.

In this proposed study, 10 patients who have symptomatic uterine adenomyosis who meet the study inclusion criteria will be invited to participate in the study which involves the use of HIFU in the management of the adenomyosis. Background information of the patients such as age, body mass index, hormonal (pre- or postmenopausal) status and the presence of chronic medical disease will be collected. Subjects will also be asked to complete an eight-item section of a Uterine Fibroid Symptom and Quality Of Life Questionnaire (UFS-QOL) and menstrual pain score which evaluate the effect of the adenomyosis on the quality of life of women.

ELIGIBILITY:
Inclusion Criteria:

* Age >40 years old, with no future childbearing plans
* Age >30 years old, who has tubal sterilization
* Significant symptoms related to adenomyosis, intractable to standard medical therapy, or patient considering radiological intervention (uterine fibroid embolization) or surgery.
* Clinical uterine size less than 20 weeks gestation
* Localized adenomyotic lesion or adenomyoma identified of less than 10 cm in diameter as judged by contrast MRI, involving only anterior or posterior uterine wall and not both.
* No laparotomy scars.
* Women should be able to give consent.

Exclusion Criteria:

* Other pelvic or uncontrolled systemic diseases
* Confirmed or suspected pregnancy
* Patients who are unable to communicate with researchers during the treatment
* Patients who are contraindicated for MRI examination
* Patients with thick abdominal wall (>5 cm, as measured by MRI)
* Presence or history of acute pelvic inflammatory disease or any pelvic malignancy
* History of lower abdominal surgery, known severe pelvic endometriosis and/ or extensive pelvic adhesion
* Presence of significant sized fibroids which may interfere with the treatment or affect the outcome measures

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-08; Primary Completion 2021-03 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Perceived symptoms change after HIFU treatment By using the menstrual pain score | The changes from baseline to post 12-month treatment will be captured
  By using the menstrual pain score for pain evaluation at each follow up (i.e. from baseline to post 1- month, post 1-month to post 3-month, post 3-month to post 6-month, post 6-month to post 12-month treatment will be captured).

SECONDARY OUTCOMES:
Perceived symptoms change after HIFU treatment By using the Uterine Fibroid Symptoms Quality Of Life Questionnaire (UFS_QOL) | The changes from baseline to post12-month treatment will be captured
  By using the Uterine Fibroid Symptoms Quality Of Life Questionnaire (UFS_QOL) for symptoms evaluation at each follow up (i.e. from baseline to post 1- month, post 1-month to post 3-month, post 3-month to post 6-month, post 6-month to post 12-month treatment will be captured)
Efficacy of HIFU in reducing the size of the adenomyotic lesion and the uterus by sonographic measurements. | The changes from baseline to post 12- month treatment will be captured
  By sonographic measurements at baseline, post 1-month, post 3-month and post 12-month treatment, the size of the adenomyotic lesion and the uterus will be evaluated by physicians.
Discomfort during procedure by using 10-cm visual analogue scale | immediate after the treatment
  By using 10-cm visual analogue scales (0 = no pain, 10 = worst pain). Women will be asked to give the pain score immediately after the HIFU treatment.
Patient satisfaction score after HIFU treatment of uterine adenomyosis | Up to 12 months
  Patients will be asked to give the satisfaction score (0= not satisfactory, 5= very satisfactory) at each follow up (i.e. post treatment 1- month, 3-month, 6-month and 12- month)
Risks and adverse effects of HIFU in the treatment of adenomyosis | Up to 12 months
  Patient will be evaluated for abnormal laboratory values and/or adverse events that are related to treatment at each follow up (i.e.post treatment 1- month, 3-month, 6-month and 12- month)
Subsequent management after HIFU treatment of uterine adenomyosis | Up to 12 months
  By physician's judgment at each follow up (i.e. at post treatment 1 months, 3 months, 6 months and 12 months), the need for subsequent additional treatments (such as hysterectomy, uterine artery embolization, or any type of hormonal treatment) will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent YT Cheung, MBBS, FRCOG, Principal Investigator — Queen Mary Hospital, Hong Kong
Locations (1):
- Hong Kong, Hong Kong